CLINICAL TRIAL: NCT05478252
Title: Investigation of Clinical Comparability of Semaglutide Drug Products Based on the Proposed and the Approved Drug Substance Manufacturing Processes in Participants With Type 2 Diabetes
Brief Title: A Research Study to Compare Two Semaglutide Medicines in People With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NN9535-4820; U1111-1266-2391 (Other: World Health Organization (WHO)); 2021-001501-69 (EudraCT Number)
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide J (Experimental): Participants will initially receive 0.25 milligrams (mg) subcutaneous injections of semaglutide J once weekly (OW) and the dose will be then escalated once in 4 weeks for 8 weeks until the target maintenance dose of 1.0 mg is reached which will be maintained for a period of 20 weeks. Metformin will be considered as background therapy during the trial.
  Interventions: Drug: Semaglutide J
- Semaglutide B (Active Comparator): Participants will initially receive 0.25 mg subcutaneous injections of semaglutide B OW and the dose will be then escalated once in 4 weeks for 8 weeks until the target maintenance dose of 1.0 mg is reached which will be maintained for a period of 20 weeks. Metformin will be considered as background therapy during the trial.
  Interventions: Drug: Semaglutide B

INTERVENTIONS:
Drug: Semaglutide J — Participants will initially receive 0.25 mg subcutaneous injections of semaglutide J OW and the dose will be then escalated once in 4 weeks for 8 weeks until the target maintenance dose of 1.0 mg is reached which will be maintained for a period of 20 weeks: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 28).
  Arms: Semaglutide J
Drug: Semaglutide B — Participants will initially receive 0.25 mg subcutaneous injections of semaglutide B OW and the dose will be then escalated once in 4 weeks for 8 weeks until the target maintenance dose of 1.0 mg is reached which will be maintained for a period of 20 weeks: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 28).
  Arms: Semaglutide B

SUMMARY:
The study compares two semaglutide medicines and looks at how well they control blood sugar levels, in participants with type 2 diabetes (T2D). Participants will either get the currently available semaglutide or the semaglutide which is produced through a new manufacturing process. Participants need to take one injection of semaglutide once a week, on the same day of every week. Participants will have a total of 11 clinic visits and the study will last for about 35 weeks (approximately 8 months).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes (T2D) mellitus greater than equal to (≥) 180 days before screening.
* Stable daily dose(s) ≥ 90 days prior to the day of screening of metformin ≥ 1500 milligrams (mg) or maximum tolerated or effective dose.
* HbA1c of 7.0-10.5 percentage (%) [53-91.3 millimoles per mole (mmol/mol)] (both inclusive).

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 days and prior insulin treatment for gestational diabetes are allowed.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for nondilated examination.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 388 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (104):
- United States (55):
  - Prime Medical Group, LLC, Gilbert, Arizona
  - FDRC, Costa Mesa, California
  - Velocity Clinical Research San Diego, La Mesa, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - LCGK Research, San Carlos, California
  - San Diego Family Care_San Diego, San Diego, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - Med Partners, Inc., Toluca Lake, California
  - University Clin Investigators, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Innovative Research of W Florida Inc., Clearwater, Florida
  - Innovative Research of W FL, Clearwater, Florida
  - Alliance for Multispec Res, Coral Gables, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - New Horizon Research Center, Miami, Florida
  - Reyes Clinical Research, Inc, Miami, Florida
  - International Research Associates, LLC_Miami, Miami, Florida
  - South Broward Research LLC, Miramar, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Omega Research Consultants LLC, Orlando, Florida
  - South Broward Research LLC, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - CVS Store Number: 7689, Atlanta, Georgia
  - CVS Store Number: 05520, Savannah, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Macoupin Research Group, Gillespie, Illinois
  - Clin Invest Spec, Inc, Wauconda, Illinois
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - MD Medical Research, Oxon Hill, Maryland
  - BTC of New Bedford, LLC, New Bedford, Massachusetts
  - Elite Research Center, Flint, Michigan
  - Arcturus Healthcare, PLC., Troy, Michigan
  - Montana Medical Research, Missoula, Montana
  - N.Y. Family Practice Physicians, Woodhaven, New York
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Whiteville Medical Assoc, PA, Whiteville, North Carolina
  - Albert J Weisbrot, Mason, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - Tristar Clin Investigations, PC, Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Elligo Clin Res Centre, Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Tapia Internal Medicine Clinic, Paris, Texas
  - Univ Of Texas Hlth Science Cntr, San Antonio, Texas
  - VIP Trials_San Antonio, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Dwayne O. Williams, M.D., P.A., Sugar Land, Texas
  - Sugar Lakes Family Practice PA, Sugar Land, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - CVS Store Number: 01396, Reston, Virginia
  - CVS Store Number: 1537, Richmond, Virginia
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
- Canada (21):
  - Care Clinic, Red Deer, Alberta
  - Ocean West Research Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Centricity Research New Minas, New Minas, Nova Scotia
  - Centricity Research Brampton, Brampton, Ontario
  - LMC Clin Res Inc. Thornhill, Concord, Ontario
  - Medical Trust Clinics, Inc., Courtice, Ontario
  - Centricity Research Etobicoke, Etobicoke, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Milestone Research, London, Ontario
  - Bluewater Clin Res Group,Inc, Sarnia, Ontario
  - Canadian Centre for Research on Diabetes_Smiths Falls, Smiths Falls, Ontario
  - LMC Endo Centres Ltd.(Bayview), Toronto, Ontario
  - LMC Manna Research, Toronto, Ontario
  - Manna Research Quebec, Lévis, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Montreal, Quebec
  - Centricity Res Pointe-Claire, Pointe-Claire, Quebec
  - Manna Research Inc., Pointe-Claire, Quebec
  - Centricity Research Ville St. Laurent VSL, Saint-Laurent, Quebec
- Poland (12):
  - Beata Miklaszewicz&Dariusz Dabrowski "CARDIAMED" s.j., Legnica, Lower Silesian Voivodeship
  - ETG Lublin, Lublin, Lublin Voivodeship
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik, Bialystok
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok
  - M2M Badania Kliniczne, Chorzów
  - NZOZ Gdanska Poradnia Cukrzycowa Sp.z o.o., Gdansk
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - FutureMeds Sp. z o.o. Lodz, Lodz
  - ETG Lublin, Lublin
  - Centrum Medyczne "Diabetika", Radom
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
  - FutureMeds Sp. z o.o., Wroclaw
- Slovakia (7):
  - Diabetologicka ambulancia DIASTYLE s.r.o., Banská Bystrica
  - Diabetologicka ambulancia DIAMO s.r.o., Kežmarok
  - IVAMEDIC s.r.o., Košice
  - DIA - SANTMART, s.r.o., Ambulancia diabetologie a poruch latkovej premeny a vyzivy, Martin
  - Diabetologicka ambulancia MUDr. Iveta Markova s.r.o, Nitra
  - MUDr. Jan Culak, s.r.o., Prievidza
  - MEDI-DIA s.r.o., Sabinov
- South Africa (9):
  - Medi-Clinic Bloemfontein, Bloemfontein, Free State
  - Moriana Clinical Research, Winnie Mandela, Free State
  - Shop#1 Health Emporium, Midrand, Gauteng
  - Prinshof Medical Campus, Pretoria, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Clinical Trial Systems (CTC), Pretoria, Gauteng
  - Dr A Amod, Durban, KwaZulu-Natal
  - Precise Clinical Solutions (Pty) Ltd, Durban, KwaZulu-Natal
  - Dr Pillay's Rooms, Durban, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 73 sites in Slovakia, Poland, South Africa, the United States and Canada.
Groups:
- Semaglutide J: Participants initially received 0.25 mg subcutaneous injections of semaglutide J once weekly and the dose was then escalated (0.25 mg in week 0 to week 4 and 0.5 mg in week 4 to week 8) once in 4 weeks until the target maintenance dose of 1.0 mg was reached which was maintained for a period of 20 weeks. Total treatment period was 28 weeks.
- Semaglutide B: Participants initially received 0.25 mg subcutaneous injections of semaglutide B once weekly and the dose was then escalated (0.25 mg in week 0 to week 4 and 0.5 mg in week 4 to week 8) once in 4 weeks until the target maintenance dose of 1.0 mg was reached which was maintained for a period of 20 weeks. Total treatment period was 28 weeks.
Period: Overall Study
Arm/Group | Semaglutide J | Semaglutide B
Started | 291 | 97
Full Analysis Set | 291 | 97
Safety Analysis Set | 291 | 97
Completed | 283 | 91
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 4 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide J | Semaglutide B | Total
Number analyzed (Participants) | 291 | 97 | 388
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (7.7) | 54.8 (7.1) | 54.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 47 | 175
  Male | 163 | 50 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 25 | 81
  Not Hispanic or Latino | 235 | 72 | 307
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 12 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 48 | 12 | 60
  White | 214 | 72 | 286
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (week 0) to end of treatment (week 28) is presented. The endpoint was evaluated based on the data from in-study period. The in-study period is defined as the uninterrupted time interval from date of randomisation to date of least contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 28)
Population: Full analysis set included all randomised participants. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 285 | 91
Percentage of glycosylated haemoglobin | -1.7 (1.0) | -1.6 (1.0)
Statistical Analysis 1: Comparison: Semaglutide J vs Semaglutide B; Test type: Non-Inferiority — Non-inferiority of insulin semaglutide J versus insulin semaglutide B was considered as confirmed if the 95% confidence interval (CI) for the mean treatment difference lied entirely below 2.5%. Non-inferiority was investigated on the FAS; p < .0001, ANCOVA; Treatment difference = -0.11, 95% CI 2-sided [-0.30 to 0.08]

2. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to end of treatment (week 28) is presented. The endpoint was evaluated based on the data from in-study period. The in-study period is defined as the uninterrupted time interval from date of randomisation to date of least contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 284 | 91
Kilogram (kg) | -5.0 (5.0) | -4.6 (4.4)

3. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of IMP, whether or not considered related to the IMP. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an IMP. All presented adverse events are TEAE. A TEAE is defined as an adverse event with an onset date (or increase in severity) during the on-treatment observation period. On-treatment observation period is defined as from first drug date until the end of study.
Time Frame: From the time of first dosing (week 0) to end of study (week 33)
Population: Safety analysis set included all participants who are exposed to study intervention.
Measure: Number; unit: Events
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 291 | 97
Events | 156 | 52

4. Secondary Outcome: Occurrence of Anti-semaglutide Antibodies (Yes/no)
Description: Occurrence of anti-semaglutide antibodies for in-study observation period is presented. The in-study period is defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. In the reported data 'yes' infers who tested positive for anti-semaglutide antibodies, whereas 'No' infers who tested negative for anti semaglutide antibodies.
Time Frame: From baseline (week 0) to end of study (week 33)
Population: Safety analysis set included all participants who are exposed to study intervention. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 282 | 90
Participants
  Yes | 1 | 0
  No | 281 | 90

5. Secondary Outcome: Occurrence of Anti-semaglutide Antibodies With In-vitro Neutralising Effect (Yes/no)
Description: Occurrence of anti-semaglutide antibodies with in-vitro neutralizing effect was to be performed based on positive cross -reactivity to GLP-1. Since there was no sample with positive cross -reactivity to GLP-1, no further analysis was performed for invitro neutralizing effect towards native-GLP1. Therefore, no data is available for this end point. In the reported data 'yes' infers who tested positive for anti-semaglutide antibodies whereas 'No' infers who tested negative for anti-semaglutide antibodies.
Time Frame: From baseline (week 0) to end of study (week 33)
Population: Since there was no sample with positive cross -reactivity to GLP-1, no further analysis was performed for invitro neutralizing effect towards native-GLP1. Therefore, no data is available for this end point.
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies Cross-reacting With Endogenous Glucagon Like Peptide-1 (GLP-1) (Yes/no)
Description: Occurrence of anti-semaglutide binding antibodies cross-reacting with endogenous glucagon like peptide-1 (GLP-1) for in-study observation period is presented. The in-study period is defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. In the reported data 'yes' infers who tested positive for anti-semaglutide binding antibodies cross-reacting with endogenous glucagon like peptide-1 (GLP-1) whereas 'No' infers who tested negative for anti-semaglutide binding antibodies cross-reacting with endogenous glucagon like peptide-1 (GLP-1).
Time Frame: From baseline (week 0) to end of study (week 33)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 1 | 0
Participants
  Yes | 0 | 0
  No | 1 | 0

7. Secondary Outcome: Occurrence of In-vitro Neutralising Cross-reacting Antibodies to Endogenous GLP-1 (Yes/no)
Description: Occurrence of in-vitro neutralising cross-reacting antibodies to endogenous GLP-1 at week 33 is presented. In the reported data 'yes' infers who tested positive for in-vitro neutralising cross-reacting antibodies to endogenous GLP-1 whereas 'No' infers who tested negative for in-vitro neutralising cross-reacting antibodies to endogenous GLP-1.
Time Frame: At week 33
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 1 | 0
Participants
  Yes | 0 | 0
  No | 1 | 0

8. Secondary Outcome: Anti-semaglutide Antibodies Level Measured as Percentage (%) Bound/Total
Description: Anti-semaglutide antibodies level measured as %Bound/Total at week 33 is presented.
Time Frame: At week 33
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of Antisemaglutide Antibodies
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 1 | 0
Percentage of Antisemaglutide Antibodies | 3.47 (0.00) |

9. Secondary Outcome: Anti-semaglutide Antibodies Level (Measured as Titre)
Description: Anti-semaglutide antibodies level measured as titre at week 33 is presented.
Time Frame: At week 33
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Titre
Arm/Group | Semaglutide J | Semaglutide B
Number analyzed (Participants) | 1 | 0
Titre | 15.00 (0.00) |

ADVERSE EVENTS:
Time Frame: From the time of first dosing (week 0) to end of study (week 33)
Description: All presented AEs are treatment-emergent (i.e., TEAEs). A TEAE is defined as an adverse event with an onset date (or increase in severity) during the on-treatment observation period. On-treatment observation period is defined as from first drug date until the end of study.
Arm/Group | Semaglutide J | Semaglutide B
All-Cause Mortality (participants affected / at risk) | 1/291 | 0/97
Serious Adverse Events (participants affected / at risk) | 8/291 | 5/97
Other Adverse Events (participants affected / at risk) | 64/291 | 24/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide J (N=291) | Semaglutide B (N=97)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide J (N=291) | Semaglutide B (N=97)
Diarrhoea (Gastrointestinal disorders) | 26 (32) | 7 (8)
Headache (Nervous system disorders) | 17 (19) | 2 (2)
Nausea (Gastrointestinal disorders) | 35 (58) | 15 (18)
Vomiting (Gastrointestinal disorders) | 15 (16) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT05478252/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT05478252/SAP_001.pdf